CLINICAL TRIAL: NCT06332586
Title: The Learning Effect of Applying Diversified Teaching in Emergency Injury Classification -Taking the Emergency Nurse of a Regional Hospital in Yunlin County as an Example
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202311087RINA
Record Dates: First submitted 2024-01-28; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-02

CONDITIONS: Triage
Keywords: Triage nurse; Diversified teaching

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The learning effect of applying diversified teaching in emergency triage and classification (Experimental)
  Interventions: Behavioral: Diversified teaching

INTERVENTIONS:
Behavioral: Diversified teaching — Diversified teaching (read and jointly mark the key points of the triage diagnosis teaching manual and read the TMS online course at any time, 1 triage diagnosis seminar/quarter, interactive teaching) for triage diagnosis nurses

SUMMARY:
"Triage" is the first process of emergency treatment. It is mainly based on the severity of the disease and the appropriate allocation of limited people, time, place, and medical resources. It is very important and related to the quality of medical care. In order to accurately judge the severity of patients, reduce the individual errors of artificial memory and increase the consistency of the judgment of triage levels, the new emergency five-level triage classification standard (Taiwan Triage and Acuity Scale) was implemented in 2010. , TTAS), the purpose is to allocate medical resources in the most appropriate manner at the appropriate time. It has been revised many times so far, so correct injury classification can maximize the safety of people's lives. This article reviews the relevant literature and finds that to have an efficient injury classification so that each patient receives appropriate medical allocation, an organized, effective and systematic injury inspection process structure is needed to enable the injury nurse to perform correct inspections. Injury skills and cognition should be actively promoted, and this policy must require traumatization nurses to continuously update their traumatization cognition and skills, and must also continue to conduct regular assessments and reviews to continuously improve the quality of traumatization grading by traumatization nurses. It can be seen that triage nurses must have skills, knowledge, attitudes and systems to improve the accuracy of triage levels and ensure the treatment of patients who need priority treatment . Therefore, this study can be used to understand the learning effectiveness of trauma care before and after diversified teaching, which can be used as a basis for teaching new trauma care nurses.

DETAILED DESCRIPTION:
On the basis of existing nursing care, in addition to improving clinical experience, trauma assessment nurses need to receive regular trauma assessment education and training, and continue to learn to gain extensive clinical cognition and skills, which can provide the best trauma assessment and classification skills; Since the triage and classification process is dynamic, situational simulations can be used to imitate real-life situations so that triage nurses can gain in-depth understanding, increase learning effects and build confidence, strengthen clinical judgment abilities, and jointly reflect and discuss to re-examine case judgment thinking. After communication, Experience records can be shared to promote improvement next time; books or structures on inspection level classification knowledge and procedures can be produced within the department and reviewed quarterly; continuous evaluation and review can be carried out to ensure the accuracy of the implemented assessment. and effectiveness, so that the triage nurse can be proficient in triage classification and decision-making, thereby improving the accuracy of triage. Therefore, triage nurses need standardized training and continuous triage education training for triage classification, which can improve the accuracy of triage. The efficiency of the injury classification by the casualty nurse also increases the self-confidence, allowing the injury nurse to perform correct injury classification more efficiently, so as to ensure that the injury classification is prioritized according to the patient's urgency and within limited resources and time. Get appropriate treatment and resource allocation within the period.

After synthesizing relevant literature, this study used the injury diagnosis judgment ability assessment test, injury diagnosis practice checklist, and satisfaction to evaluate the learning effectiveness before using diversified teaching. While using diversified teaching (reading and jointly marking the key points of the trauma diagnosis teaching manual and reading TMS online courses at any time, trauma examination seminar once/quarter, interactive teaching) for trauma examination nurses, using the trauma assessment judgment ability assessment test, Injury diagnosis practice checklist and satisfaction assessment of learning effectiveness.

The subjects of the study were emergency trauma nurses, and the purpose and method of the research, as well as informed consent, were explained to them. The emergency nurses filled out a questionnaire and informed consent form during their break. The content included basic information and case scenario simulation assessments, and through trauma examination The instructor randomly conducts daily field audits in three shifts (12 times/month), collects and archives all questionnaire data, and then conducts statistical analysis with SPSS version 25. The research results belong to National Taiwan University Hospital, and the results may be published in academic papers and other applications in the future.

ELIGIBILITY:
Inclusion Criteria:

* Pass Nursing Advanced 2
* New medical examiner

Exclusion Criteria:

* Nursing advanced level has not reached advanced level 2
* Not a new review nurse

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-03-25 (Estimated); Primary Completion 2024-04-04 (Estimated); Study Completion 2024-05-05 (Estimated)

PRIMARY OUTCOMES:
Improving the injury diagnosis ability of triage diagnosis nurses through diversified teaching | six week
  Use diversified teaching to improve the ability of triage diagnosis nurses

CONTACTS AND LOCATIONS:
Locations (1):
- Taiwan, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] AlShatarat M, Rayan A, Eshah NF, Baqeas MH, Jaber MJ, ALBashtawy M. Triage Knowledge and Practice and Associated Factors Among Emergency Department Nurses. SAGE Open Nurs. 2022 Oct 3;8:23779608221130588. doi: 10.1177/23779608221130588. eCollection 2022 Jan-Dec. PMID 36213615
- See also: Triage Knowledge and Practice and Associated Factors Among Emergency Department Nurses — https://pubmed.ncbi.nlm.nih.gov/36213615/